CLINICAL TRIAL: NCT01231399
Title: Phase Ib Trial of mFOLFOX6 and Everolimus (NSC-733504) in Patients With Metastatic Gastroesophageal Adenocarcinoma
Brief Title: Everolimus and Combination Chemotherapy in Treating Patients With Metastatic Stomach or Esophageal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10064; NCI-2010-02168
Record Dates: First submitted 2010-10-28; First posted 2010-11-01 (Estimated); Results first posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-04

CONDITIONS: Adenocarcinoma of the Esophagus; Adenocarcinoma of the Gastroesophageal Junction; Diffuse Adenocarcinoma of the Stomach; Intestinal Adenocarcinoma of the Stomach; Mixed Adenocarcinoma of the Stomach; Recurrent Esophageal Cancer; Recurrent Gastric Cancer; Stage IV Esophageal Cancer; Stage IV Gastric Cancer
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Neoplasms; Stomach Neoplasms | interventions — Fluorouracil; Leucovorin; Oxaliplatin; Everolimus; Immunohistochemistry; Microarray Analysis; Gene Expression Profiling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients receive fluorouracil IV continuously over 46 hours, leucovorin calcium IV over 2 hours, and oxaliplatin IV over 2 hours on day 1. Patients also receive oral everolimus once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin; Drug: everolimus; Other: laboratory biomarker analysis; Other: immunohistochemistry staining method; Genetic: microarray analysis

INTERVENTIONS:
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU; Adrucil; Efudex; FU
Drug: leucovorin calcium — Given IV
  Other Names: calcium folinate; CF; CFR; citrovorum factor; LV; Wellcovorin
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; diaminocyclohexane oxalatoplatinum; Eloxatin; L-OHP
Drug: everolimus — Given orally
  Other Names: 42-O-(2-hydroxy)ethyl rapamycin; Afinitor; RAD001
Other: laboratory biomarker analysis — Correlative studies
Other: immunohistochemistry staining method — Correlative studies
  Other Names: immunohistochemistry
Genetic: microarray analysis — Correlative studies
  Other Names: gene expression profiling

SUMMARY:
RATIONALE: Everolimus may stop the growth of stomach or esophageal cancer by blocking blood flow to the tumor. Drugs used in chemotherapy, such as leucovorin calcium, fluorouracil, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing, or by stopping them from spreading. Giving everolimus together with combination chemotherapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of everolimus when given together with combination chemotherapy in treating patients with metastatic stomach or esophageal cancer that has spread to other places in the body.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To determine the maximum tolerated dose of everolimus to use in combination with mFOLFOX6 [oxaliplatin, leucovorin (leucovorin calcium), 5-FU (fluorouracil)].

II. To better describe the toxicities associated with the combination of everolimus with mFOLFOX6.

III. To assess response rate and progression-free survival in this patient population.

IV. To assess overall survival in patients with metastatic gastric, esophageal and gastroesophageal junction (GEJ) adenocarcinoma treated with the combination of mFOLFOX6 + everolimus.

OUTLINE: This is a dose-escalation study of everolimus. Patients receive fluorouracil intravenously (IV) continuously over 46 hours, leucovorin calcium IV over 2 hours, and oxaliplatin IV over 2 hours on day 1. Patients also receive oral everolimus once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diagnosis of gastric, esophageal, and GEJ adenocarcinoma
* Patients must have metastatic disease
* Patients must not have received any chemotherapy for metastatic disease
* Patients may have received prior adjuvant chemotherapy; completion of chemotherapy must be greater than 6 months from date of recurrent disease
* Patients must have computed tomography (CT) or magnetic resonance imaging (MRI) scan; patients must have at least one measurable site of disease according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria that has not been previously irradiated; if the patient has had previous radiation to the marker lesion(s), there must be evidence of progression since the radiation
* Patients must have a ECOG Performance Status of 0-1
* Absolute neutrophil count (ANC) > 1,500/mcl
* Platelet count > 100,000/mcl
* Hemoglobin (Hg) > 9 g/dL
* Serum creatinine < 1.5 mg/dl and/or Creatinine clearance > 60 cc/min
* Bilirubin < 1.5 mg/dl
* Serum glutamic oxaloacetic transaminase (SGOT) and/or serum glutamic pyruvic transaminase (SGPT) =< 2.5 x institutional upper limit of normal (IULN) (=< 5 x upper limit of normal [ULN] in patients with liver metastases)
* Fasting serum cholesterol =< 300 mg/dL or =< 7.75 mmol/L
* Fasting triglycerides =< 2.5 x ULN; NOTE: in case one or both of these thresholds are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication
* Patients should have controlled diabetes as evidenced by hemoglobin (Hb)A1C =< 8%
* International normalized ratio (INR) and partial thromboplastin time (PTT) =< 1.5; (anticoagulation is allowed if target INR =< 1.5 on a stable dose of warfarin or on a stable dose of low molecular weight [LMW] heparin for > 2 weeks at time of randomization)
* Due to the possibility of harm to a fetus or nursing infant from this treatment regimen, patients must not be pregnant or nursing (or plan to become pregnant); women and men of reproductive potential must have agreed to use a highly effective contraceptive method for at least 8 weeks after treatment
* Patients with risk factors for contraction hepatitis B or C should undergo screening prior to treatment on protocol. Patients with detectable viral titers are required to receive treatment for 4 weeks prior to starting protocol therapy.
* Patients must be able to swallow pills
* No other prior malignancy within the past 3 years is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* Patients must have pathology specimen available for submission

Exclusion Criteria:

* Patients currently receiving anticancer therapies or who have received anticancer therapies within 4 weeks of the start of study drug (including chemotherapy, radiation therapy, antibody based therapy, etc)
* Patients who have received prior treatment with an mammalian target of rapamycin (mTOR) inhibitor (sirolimus, temsirolimus, everolimus)
* Patients with a known hypersensitivity to everolimus or other rapamycins (sirolimus, temsirolimus) or to its excipients
* Patients, who have had a major surgery or significant traumatic injury within 4 weeks of start of study drug, patients who have not recovered from the side effects of any major surgery (defined as requiring general anesthesia) or patients that may require major surgery during the course of the study
* Prior treatment with any investigational drug within the preceding 4 weeks
* Patients receiving chronic, systemic treatment with corticosteroids (prednisone > 10 mg per day) or another immunosuppressive agent; topical or inhaled corticosteroids are allowed
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

  * Symptomatic congestive heart failure of New York heart Association Class III or IV
  * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction within 6 months of start of study drug, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease
  * Severely impaired lung function as defined as spirometry and diffusion lung capacity of carbon monoxide (DLCO) that is 50% of the normal predicted value and/or 02 saturation that is 88% or less at rest on room air
  * Uncontrolled diabetes as defined by fasting serum glucose > 1.5 x ULN
  * Active (acute or chronic) or uncontrolled severe infections
  * Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
* A known history of human immunodeficiency virus (HIV) seropositivity
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
* Patients with an active, bleeding diathesis; history of noncompliance to medical regimens
* Patients unwilling to or unable to comply with the protocol

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Chung, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - City of Hope Medical Center, Duarte, California
  - South Pasadena Cancer Center, South Pasadena, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1 - 2.5 mg Everolimus Daily: Patients receive 400 mg/m^2 fluorouracil (5-FU) IV slow push day 1, 2,400 mg/m^2 fluorouracil (5-FU) IV continuously over 46 hours days 1-2, 400 mg/m^2 leucovorin calcium IV over 2 hours, and 85 mg/m^2 oxaliplatin IV over 2 hours on day 1. Patients also receive 2.5 mg oral everolimus once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  fluorouracil: Given IV
  leucovorin calcium: Given IV
  oxaliplatin: Given IV
  everolimus: Given orally
Period: Overall Study
Arm/Group | Dose Level 1 - 2.5 mg Everolimus Daily
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dose Level 1 - 2.5 mg Everolimus Daily
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 58 [36 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Everolimus
Description: The highest dose tested in which fewer than 33% of patients experience an attributable DLT to the study drug, when at least 6 patients are treated at that dose and are evaluable for toxicity. Toxicities will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) v4.0.
Time Frame: Course 1 (first 28 days)
Population: All patients observed for 28 days while receiving a full course of therapy or who experienced a DLT. Patients withdrawing before completion of the first course, for reasons other than DLT, were replaced.
Measure: Number; unit: mg
Groups:
- Dose Level 1 - 2.5 mg Everolimus: Patients receive 400 mg/m^2 fluorouracil (5-FU) IV slow push day 1, 2,400 mg/m^2 fluorouracil (5-FU) IV continuously over 46 hours days 1-2, 400 mg/m^2 leucovorin calcium IV over 2 hours, and 85 mg/m^2 oxaliplatin IV over 2 hours on day 1. Patients also receive 2.5 mg oral everolimus once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  fluorouracil: Given IV
  leucovorin calcium: Given IV
  oxaliplatin: Given IV
  everolimus: Given orally
Arm/Group | Dose Level 1 - 2.5 mg Everolimus
Number analyzed (Participants) | 6
mg | 2.5

2. Primary Outcome: Number of Subject With Overall Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 5 years
Measure: Number; unit: participants
Arm/Group | Dose Level 1 - 2.5 mg Everolimus Daily
Number analyzed (Participants) | 6
participants | 5

3. Primary Outcome: Progression-free Survival
Description: Estimated using the product-limit method of Kaplan and Meier. From the date treatment started until the date of first documented progression or date of death from any cause, whichever came first. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: up to 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose Level 1 - 2.5 mg Everolimus Daily
Number analyzed (Participants) | 6
Months | 14.5 [2.0 to 21.0]

4. Primary Outcome: Overall Survival
Description: Estimated using the product-limit method of Kaplan and Meier. From the date treatment started until the date of death from any cause.
Time Frame: Up to 5 years.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose Level 1 - 2.5 mg Everolimus Daily
Number analyzed (Participants) | 6
Months | 20.3 [15.6 to 28.9]

ADVERSE EVENTS:
Time Frame: Adverse events occurred over a period of 2 years, 6 months
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Dose Level 1 - 2.5 mg Everolimus Daily
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 - 2.5 mg Everolimus Daily (N=6)
Mucositis oral (Gastrointestinal disorders) | 1 (2)
Chills (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 - 2.5 mg Everolimus Daily (N=6)
Hyperglycemia (Investigations) | 4 (8)
Hypocalcemia (Investigations) | 3 (15)
Anemia (Blood and lymphatic system disorders) | 6 (66)
Sinus bradycardia (Cardiac disorders) | 2 (5)
Sinus tachycardia (Cardiac disorders) | 3 (8)
Watering eyes (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (25)
Bloating (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (21)
Diarrhea (Gastrointestinal disorders) | 3 (6)
Dry mouth (Gastrointestinal disorders) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 3 (6)
Dysphagia (Gastrointestinal disorders) | 2 (5)
Esophageal pain (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (9)
Gastrointestinal disorders - Other, spec (Gastrointestinal disorders) | 2 (3)
Hemorrhoids (Gastrointestinal disorders) | 1 (3)
Mucositis oral (Gastrointestinal disorders) | 4 (14)
Nausea (Gastrointestinal disorders) | 6 (34)
Oral pain (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 3 (5)
Chills (General disorders) | 1 (2)
Edema face (General disorders) | 1 (1)
Fatigue (General disorders) | 6 (56)
Fever (General disorders) | 2 (4)
Flu like symptoms (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Injection site reaction (General disorders) | 2 (3)
Pain (General disorders) | 2 (4)
Mucosal infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (3)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Activated partial thromboplastin time pr (Investigations) | 2 (10)
Alanine aminotransferase increased (Investigations) | 5 (31)
Alkaline phosphatase increased (Investigations) | 5 (35)
Aspartate aminotransferase increased (Investigations) | 5 (37)
CPK increased (Investigations) | 1 (2)
Cholesterol high (Investigations) | 5 (32)
Creatinine increased (Investigations) | 1 (2)
Haptoglobin decreased (Investigations) | 1 (1)
INR increased (Investigations) | 1 (8)
Lymphocyte count decreased (Investigations) | 3 (8)
Lymphocyte count increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 6 (29)
Platelet count decreased (Investigations) | 5 (30)
Weight gain (Investigations) | 2 (3)
Weight loss (Investigations) | 3 (17)
White blood cell decreased (Investigations) | 6 (28)
Anorexia (Metabolism and nutrition disorders) | 4 (17)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 4 (37)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (11)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 3 (19)
Obesity (Metabolism and nutrition disorders) | 3 (17)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (20)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue di (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (5)
Akathisia (Nervous system disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (2)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 3 (10)
Dysphasia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Memory impairment (Nervous system disorders) | 1 (2)
Paresthesia (Nervous system disorders) | 4 (12)
Peripheral motor neuropathy (Nervous system disorders) | 2 (6)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (30)
Somnolence (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (13)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (11)
Confusion (Psychiatric disorders) | 2 (3)
Depression (Psychiatric disorders) | 3 (20)
Insomnia (Psychiatric disorders) | 2 (23)
Restlessness (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 3 (11)
Proteinuria (Renal and urinary disorders) | 3 (9)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal di (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (9)
Skin and subcutaneous tissue disorders - (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 6 (74)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes